CLINICAL TRIAL: NCT07143188
Title: Elemental Diet as an Adjunctive Therapy for Inflammatory Bowel Disease Flares The EDICT Trial
Brief Title: The EDICT Trial - Therapy for Inflammatory Bowel Disease Flares
Acronym: EDICT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: mBIOTA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00126650
Record Dates: First submitted 2025-08-19; First posted 2025-08-27 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-08

CONDITIONS: Inflammatory Bowel Disease
Keywords: crohn's disease; ulcerative colitis; chronic gastrointestinal tract inflammation
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — Food, Formulated

STUDY DESIGN:
Intervention Model Description: randomized, open-label, parallel group controlled trial - Patients with an established diagnosis of Inflammatory bowel disease (Crohn's disease (CD) or ulcerative colitis (UC)) who are having a flare will be assessed for eligibility criteria; eligible patients will be randomized to one of two groups, both of which will receive standard of care pharmacologic treatment: 1) a control group which will receive standard dietary advice; 2) a treatment group in which all nutrition will be provided by mBIOTA elemental diet for 2 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- elemental diet (ED) (Experimental): The intervention in this study will be an elemental diet (ED) formulation produced by mBIOTA. All patients randomized to the ED arm will receive a two-week supply (84 servings + additional packets as needed) of the "original" flavor mBIOTA elemental diet.
  Interventions: Dietary Supplement: elemental diet (ED)
- control group (No Intervention): Patients randomized to the control group will undergo counseling with a registered dietician for general dietary advice but will be instructed to continue their usual diet, as tolerated, without any restrictions.

INTERVENTIONS:
Dietary Supplement: elemental diet (ED) — mBIOTA is a palatable elemental diet formulation
  Other Names: mBIOTA elemental diet
  Arms: elemental diet (ED)

SUMMARY:
Inflammatory bowel disease (IBD), including Crohn's disease (CD) and ulcerative colitis (UC), are chronic inflammatory conditions of the gastrointestinal tract that affect millions of people in the United States of America. Among patients with IBD, symptomatic flares are quite common; up to 40-50% of patients in some populations report having a flare at least once per month. For most patients with IBD flares, the typical outpatient treatment consists of corticosteroids and, in some instances, initiation of or switching between 5-aminosalicylic acid-acid preparations, immunomodulators, or biologics. These treatments, while often effective, can have harmful side effects, especially when used for long durations of time. Therefore, alternative treatments are highly sought after by both patients and providers.

DETAILED DESCRIPTION:
Enteral nutrition (EN) has shown promise in treating IBD and has the theoretical benefit of reducing symptoms and increasing quality of life while avoiding the side effects associated with standard pharmacotherapy. Exclusive EN has even proven superior to steroids for induction of remission in CD in pediatric patients. Unfortunately, the same effect has not been seen in adults, but a Chochrane metaanalysis showed no significant difference in remission rates between steroids and exclusive EN for treatment of CD. Notably, however, EN studies are notoriously hindered by small group sizes and limited adherence to study diets due to poor palatability. Therefore, although exclusive EN may have a role in IBD treatment, there is limited data to support its use.

Elemental diets (ED) are a form of enteral nutrition in which free amino acids, mono- and polysaccharides, short or medium chain triglycerides, vitamins, and minerals are combined to provide a complete nutritional source. EDs have a long history of use in treating inflammatory diseases of the GI tract, such as IBD, eosinophilic esophagitis, and small intestinal bacterial overgrowth. The hypothesized benefit of EDs stems from their highly efficient absorption that requires minimal digestion, as well as the absence of allergenic antigens. As with other EN studies, examining the use of EDs for treatment of inflammatory gastrointestinal diseases have been limited by very poor palatability.

mBIOTA is a palatable elemental diet formulation that may be a more acceptable treatment option for a variety of GI problems. In a head-to-head comparison survey, mBIOTA outperformed its leading market competitor in six palatability domains (taste, smell, consistency, aftertaste, appearance, and impression). In a recently published study investigating ED for treatment of small intestinal bacterial overgrowth, subjects had a 100% adherence rate to mBIOTA supplementation during the trial period. Given its improved palatability compared to its predecessors, mBIOTA could prove useful as a new therapeutic tool in the treatment of inflammatory bowel disease.

ELIGIBILITY:
Inclusion Criteria:

* adults with an established diagnosis of inflammatory bowel disease (ulcerative colitis or Crohn's disease) who are being treated in the outpatient setting for an Inflammatory bowel disease (IBD) flare, defined as a clinically significant increase in IBD symptoms (e.g., abdominal pain, nausea, vomiting, diarrhea, joint pain, fever, bleeding, unintended weight loss).

Exclusion Criteria:

* Patients requiring admission to the hospital for treatment of a flare
* Patients with allergies to any ingredients in the mBIOTA Elemental Diet
* Female patients who are pregnant
* Patients with diabetes who are taking insulin as part of their treatment plan
* Patients with other medical conditions or personal preferences that would compromise their ability to adhere to the elemental study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
change of symptom burden scores | Week 1 to Week 12
  assessed by the symptom severity survey - collecting all data using the same survey for both Crohn's disease and ulcerative colitis patients.
  the Simple Clinical Colitis Activity Index (SCCAI) ranges from 0-19. For both scores, lower means less disease activity and therefore "better." the Harvey-Bradshaw Index (HBI) - Based on convention, a total HBI score of <5 indicates remission, 5-7 suggests mild severity, 8-16 denotes moderate severity, and ≥16 demarks severe disease.

SECONDARY OUTCOMES:
changes in inflammatory markers - Erythrocyte Sedimentation Rate (ESR) | Baseline, Weeks 2 and 4
  a blood test that measures the rate at which red blood cells settle at the bottom of a test tube. This rate is an indicator of inflammation in the body, with a faster settling rate suggesting higher inflammation. It's a general marker, meaning it can be elevated in various conditions, but it's not specific to any single disease - High ESR: Suggests inflammation, which could be due to infections, autoimmune diseases, or some types of cancer.
  Normal ESR: Doesn't always rule out inflammation, as some inflammatory conditions may not cause a significant ESR elevation.
changes in inflammatory markers - C-reactive protein (CRP) | Baseline, Weeks 2 and 4
  a blood test that measures inflammation in the body. It's an acute-phase reactant, meaning its levels rise in response to inflammation or infection. Elevated CRP can indicate various conditions, including infections, autoimmune diseases, and even heart disease risk.
  Normal:
  Generally, a level below 1.0 mg/dL is considered normal, according to the National Institutes of Health (NIH).
  Mildly elevated:
  Levels between 1.0 and 10.0 mg/dL may indicate conditions like obesity, pregnancy, or minor infections.
  Moderately elevated:
  Levels between 10.0 and 100.0 mg/dL can be associated with autoimmune diseases, pancreatitis, or bronchitis.
  Markedly elevated:
  Levels above 100.0 mg/dL often suggest acute bacterial infection, major trauma, or severe inflammation.
changes in inflammatory markers - fecal calprotectin | Baseline, Weeks 2 and 4
  a valuable inflammatory marker, particularly for assessing gastrointestinal inflammation, and is often used in the diagnosis and management of inflammatory bowel disease (IBD). It is a protein released by neutrophils (white blood cells) that are recruited to sites of inflammation in the gut. Elevated levels of fecal calprotectin suggest active inflammation in the intestines.
changes in nutritional status - Prealbumin | Baseline, Weeks 2 and 4
  Prealbumin is a measure of nutritional status, with a low level meaning undernutrition. The normal range is 15-36 Low levels (<15 mg/dL) may indicate malnutrition, protein deficiency, inflammation, or liver disease.
  High levels (>36 mg/dL) may be seen in certain medications (e.g., corticosteroids), kidney failure, or multiple myeloma.
changes in nutritional status - Bioelectrical Impedance Analysis score | Baseline, Weeks 2 and 4
  Bioelectrical Impedance Analysis score (BIA) will be used to estimate lean muscle mass (body cell mass) and fat mass. Ideal body cell mass in men is estimated as 40-45% of ideal body weight for height. For women, the ideal body cell mass is estimated at 30-35% of ideal body weight for height. Ideal fat mass for men is around 10-20% of actual body weight. Ideal fat mass for women is estimated at 20-30% of actual body weight.
number of prednisone equivalents | Week 12
  total amount of supplemental steroids given as treatment of inflammatory bowel disease, measured as prednisone equivalents
number of Emergency Department visits or hospitalization visits | Week 1 to Week 12
  number of Emergency Department visits or hospitalization visits

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Weinberg, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No